CLINICAL TRIAL: NCT03402984
Title: Acotiamide Affects Antral Motility, But Has no Effect on Fundic Motility, Gastric Emptying or Symptom Perception in Healthy Participants
Brief Title: Effect of Acotiamide on Gastric Motility and Satiation in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: Acotiamide1
Record Dates: First submitted 2018-01-10; First posted 2018-01-18 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Healthy
Keywords: Gastric motility; Gastric emptying
MeSH Terms: interventions — Z 338

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acotiamide (Experimental): Acotiamide 100 mg t.i.d. for 3 weeks. Intake of medication 10 minutes before meal.
  Interventions: Drug: Acotiamide
- Placebo (Placebo Comparator): Placebo tablets, t.i.d. for 3 weeks. Intake of placebo 10 minutes before meal.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Acotiamide — Acotiamide treatment, 100 mg, t.i.d. for three week. Intake 10 minutes before meal.
  Arms: Acotiamide
Drug: Placebo Oral Tablet — Placebo treatment, t.i.d. for three week. Intake 10 minutes before meal.
  Arms: Placebo

SUMMARY:
Introduction. Functional dyspepsia (FD) is a common chronic gastrointestinal disorder with a high socio-economic impact. Acotiamide, a new prokinetic agent, was shown to be efficacious in the treatment of FD, especially in the postprandial distress syndrome subgroup. To date, the exact mechanism of action of acotiamide is incompletely elucidated.

The aim of this study was to examine the effect of acotiamide on gastric motility, gastric emptying rate and gastrointestinal symptom perception in healthy participants in a randomized, placebo-controlled, cross-over study design. Participants were treated with acotiamide (100 mg t.i.d.) and placebo for 3 weeks, separated by a one-week wash-out period. At the end of each treatment period, gastric emptying and motility were assessed on two consecutive study days. During gastric motility assessment, epigastric symptom scores were collected at multiple time points.

ELIGIBILITY:
Inclusion Criteria:

* age: 18-60 years old.
* Participant must provide witnessed written informed consent prior to any study procedures being performed.

Exclusion criteria:

* Age > 60 years old.
* severely decreased kidney function.
* severely decreased liver function.
* severe heart disease, for example a history of irregular heartbeats, angina or heart attack.
* severe lung disease.
* severe psychiatric illness or neurological illness.
* any gastrointestinal disease.
* any dyspeptic symptoms.
* pregnant or breastfeeding.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2017-12-04 (Actual)

PRIMARY OUTCOMES:
Gastric accommodation | Gastric pressure was measured until 1 hour after the start of the liquid meal. Liquid meal started 10 minutes after medication/placebo intake
  Relaxation of the stomach upon food intake

SECONDARY OUTCOMES:
Gastric emptying | Breath samples were collected before intake of medication/placebo and every 15 minutes until 4h after intake of 13C-octanoid acid
  Gastric emptying was assess by a 13C-octanoid acid breath test
Change in subjective gastrointestinal symptom scores measured by visual analogue scale of 100 mm | assessment by questionnaire (100 mm Visual Analogue Scale) every 5 minutes, up to 1 hour after administration of the liquid meal

CONTACTS AND LOCATIONS:
Overall Officials: Jan Tack, PhD, MD, Principal Investigator — UZ Leuven / KU Leuven
Locations (1):
- Jan Tack, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Masuy I, Tack J, Verbeke K, Carbone F. Acotiamide affects antral motility, but has no effect on fundic motility, gastric emptying or symptom perception in healthy participants. Neurogastroenterol Motil. 2019 Apr;31(4):e13540. doi: 10.1111/nmo.13540. Epub 2019 Jan 20. PMID 30663175